CLINICAL TRIAL: NCT06819332
Title: An Observational Study of Pedal Cycle Related Trauma at the Royal London Hospital
Brief Title: Pedal Cycle Related Trauma at the Royal London Hospital
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 158400
Record Dates: First submitted 2017-04-19; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Bicycle Accident

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bespoke is an observational, prospective, cohort study. The aim of this study is to explore injury patterns of patients who require admission to the Royal London Hospital (RLH) Emergency Department (ED)or outpatient clinics as a result of any collision involving a bicycle. Secondary objectives are to determine the circumstances around cycling injury and to explore the effect of cycling collisions on the return to work, activities of daily living and cycling. All patients that attend the Emergency Department of the Royal London Hospital following an injury sustained while cycling, will be invited to take part in the study. Participants will be asked to answer a questionnaire about their cycling routines as well as provide information about the location, conditions and events surrounding their collision. Patients' recovery will be followed by the study team using the electronic health record and by reviewing the patients' notes. Morbidity and mortality data will be completed at death, discharge or 28 days from admission (whichever comes first). The patients will be followed up in person, email, or via telephone at 6 weeks following their initial admission. The research team hosted a Patient and Public Involvement (PPI) event, to determine which outcome measures were important for the public to investigate. It was found that the majority of the group felt it was important to follow up return to work, return to cycling and return to activities of daily living in any patients who have had a cycling collision. These outcomes will be measured at the 6 week follow up.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are 16 years and older attending the Royal London Hospital Emergency department who have been injured while riding a bicycle (pedal cycle)
* All patients who are 16 years and older who are transferred to the Royal London Hospital, either for inpatient or outpatient care, who were injured whilst riding a bicycle

Exclusion Criteria:

* Patients who have been injured while involved in activities other than cycling
* Patients that decline to take part in the study
* Patients who are 15 years or younger
* Off road cyclists
* motorbike riders

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who attend the Royal London HOSPT
Sampling Method: Non-Probability Sample
Enrollment: 644 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Epidemiology of bicycle related accidents in London in patients who present to the Royal London Hospital. | 14 days
  Measure epidemiology of bicycle related accidents in London

SECONDARY OUTCOMES:
To map collision hotspots in London and quantify and draw patients' quality of life after injury using using EQ-5D - EuroQol as a measuring tool to assess patient generic health status and SF-12 to measure functional health and well-being. | 6 Weeks (+/-2 weeks)
  Using EQ-5D - EuroQol as a measuring tool to assess patient generic health. 5-level EQ-5D version by EuroQol for descriptive and visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided